CLINICAL TRIAL: NCT03608436
Title: RECOVER Study: the Effect of Low- Versus Normal Pressure Pneumoperitoneum During Laparoscopic Colorectal Surgery on the Early Quality of Recovery With Perioperative Care According to the Enhanced Recovery Principles
Brief Title: The Effect of Low Pressure Pneumoperitoneum During Laparoscopic Colorectal Surgery on Early Quality of Recovery
Acronym: RECOVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL65290.091.18
Record Dates: First submitted 2018-06-18; First posted 2018-08-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-03

CONDITIONS: Pneumoperitoneum; Neuromuscular Blockade; Surgery
Keywords: Quality of recovery; Laparoscopic surgery; Deep neuromuscular block; Low pressure pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low pressure PNP, deep NMB (Experimental): Low pressure pneumoperitoneum of 8 mmHg with deep neuromuscular block (post tetanic count of 1-2) reached by titration with continuous infusion of Rocuronium bromide.
  Interventions: Procedure: Low pressure pneumoperitoneum; Drug: Rocuronium Bromide
- Normal pressure PNP, moderate NMB (Active Comparator): Normal pressure pneumoperitoneum of 12 mmHg with moderate neuromuscular block (TOF count of 1-2) reached by titration with bolus or continuous infusion of a low dose of Rocuronium bromide.
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Procedure: Low pressure pneumoperitoneum — Lowering intra-abdominal pressure during laparoscopic surgery
  Other Names: Low intra-abdominal pressure
  Arms: Low pressure PNP, deep NMB
Drug: Rocuronium Bromide — Deep (PTC 1-2) versus moderate (Tof count 1-2) neuromuscular block
  Other Names: Deep muscle relaxation

SUMMARY:
Randomised controlled trial comparing the effect of low pressure pneumoperitoneum with deep neuromuscular block versus normal pressure pneumoperitoneum with moderate neuromuscular block during laparoscopic colorectal surgery on early quality of recovery.

DETAILED DESCRIPTION:
Rationale: the laparoscopic approach reduced trauma as compared to open surgery, however, the pressure used to create a PNP with sufficient surgical workspace still leads to significant tissue injury. Prior studies show that the use of low-pressure pneumoperitoneum (PNP) during laparoscopic surgery reduced postoperative pain scores, cumulative opioid consumption and improved bowel function recovery. Deep neuromuscular blockade (NMB) as compared to moderate NMB decreases the amount of intra-abdominal pressure required to achieve similar surgical conditions and enables the use of low-pressure PNP without compromising the quality of the surgical field and patient safety. Therefore, the use of deep NMB with low-pressure PNP could be a significant addition to the conventional Enhanced Recovery After Surgery (ERAS) protocols.

Objective: to establish the relationship between the use of low pressure pneumoperitoneum with deep neuromuscular blockade and the early quality of recovery after laparoscopic colorectal surgery.

Study design: a multi-center, blinded, randomized controlled clinical trial.

Study population: adult individuals scheduled for laparoscopic colorectal surgery with a primary colonic anastomosis.

Intervention: participants will be randomly assigned in a 1:1 fashion to either the experimental group (group A): low pressure PNP (8 mmHg) with deep NMB (PTC 1-2) or the control group (group B): normal pressure PNP (12 mmHg) with moderate NMB (TOF count 1-2).

Primary endpoint: Quality of recovery score (QoR-40) 24 hours after surgery.

Secondary endpoints: QoR-40 score (day 3 and 7 after surgery), McGill pain- and RAND-36 score (1 day before and 3 months after surgery), pain scores, PONV, analgesia use, length of hospital stay, postoperative complications, surgical conditions and time to reach discharge criteria.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic colorectal surgery with a primary anastomosis
* Obtained informed consent
* Age over 18 years

Exclusion Criteria:

* Insufficient control of the Dutch language to read the patient information and to fill out the questionnaires
* Primary colostomy
* Neo-adjuvant chemotherapy
* Chronic use of analgesics or psychotropic drugs
* Use of NSAIDs shorter than 5 days before surgery
* Known or suspected allergy to rocuronium of sugammadex
* Neuromuscular disease
* Indication for rapid sequence induction
* Severe liver- or renal disease (creatinine clearance <30ml/min)
* BMI >35 kg/m²
* Deficiency of vitamin K dependent clotting factors or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Total score on the Quality of Recovery-40 questionnaire | 24 hours after surgery
  The QoR-40 is a validated assessment tool for measuring a patient's self-assessed quality of recovery after surgery. It consists of 40 questions measuring 5 dimensions: patient support, comfort, emotions, physical independence and pain. Each item is rated on a scale of 1 to 5, giving a minimal score of 40 and a maximum score of 200.

SECONDARY OUTCOMES:
Total score on the Quality of Recovery-40 questionnaire | Day 3 and day 7 after surgery
  The QoR-40 is a validated assessment tool for measuring a patient's self-assessed quality of recovery after surgery. It consists of 40 questions measuring 5 dimensions: patient support, comfort, emotions, physical independence and pain. Each item is rated on a scale of 1 to 5, giving a minimal score of 40 and a maximum score of 200.
McGill pain Questionnaire | Upon admission and 3 months after surgery
  Validated questionnaire for the assessment of quality and intensity of pain
RAND-36 general health questionnaire | Upon admission and 3 months after surgery
  Validated patient-reported survey of health
Pain scores | 1, 8, 24, and 72 hours after surgery
  Pain at rest and pain upon movement (NRS 0-10), is pain acceptable yes or no, referred shoulder pain yes or no?
Post-operative nausea and vomiting (PONV) | 1, 8, 24 and 72 hours after surgery
  NRS 0-10
Cumulative use of analgesics and anti-emetics | 1, 8, 24 and 72 hours after surgery
  Total dose of opiates, other analgesics and anti-emetic drugs
Length of hospital stay | From date of admission until date of discharge from the hospital (usually several days), assessed up to 3 months.
  Total number of days from admission to discharge after surgery (not including readmission)
Surgical conditions | Intraoperative: after introduction of the trocars and every 15 minutes until the end of the pneumoperitoneum.
  Rating of the surgical conditions with the Leiden Surgical Rating Scale (L-SRS). The L-SRS is scored by the surgeon and ranges from 1-5 for quality of the surgical field. A score of 5 means optimal conditions: a wide laparoscopic field with no patient movements or muscle contractions, 1 means extremely poor conditions: the surgeon is unable to obtain a visible laparoscopic field because of inadequate muscle relaxation.
Intraoperative complications | During surgery
  Complications during surgery graded according to the Clavien-Dindo classification
Postoperative complications | Up to 3 months after surgery
  Postoperative complications
Time to reach discharge criteria | From date of surgery until date of actual discharge from the hospital (usually several days), assessed up to 3 months.
  Number of days to reach the following criteria after surgery: adequate pain control with oral medication, passage of flatus or defecation, intake of solid food tolerated, patient is mobilized and independent and patient accepts discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kim I Albers, MD, Principal Investigator — Radboud University Medical Center; Michiel C Warlé, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Martini general hospital, Groningen
  - Maxima Medisch Centrum, Veldhoven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albers KI, Polat F, Panhuizen IF, Snoeck MMJ, Scheffer GJ, de Boer HD, Warle MC. The effect of low- versus normal-pressure pneumoperitoneum during laparoscopic colorectal surgery on the early quality of recovery with perioperative care according to the enhanced recovery principles (RECOVER): study protocol for a randomized controlled study. Trials. 2020 Jun 17;21(1):541. doi: 10.1186/s13063-020-04496-8. PMID 32552782